CLINICAL TRIAL: NCT00000874
Title: A Pilot Study of the Short-Term Effects of Antiretroviral Management Based on Plasma Genotypic Antiretroviral Resistance Testing (GART) Compared With Antiretroviral Management Without Plasma GART
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: CPCRA 046; 11598 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2013-10-01 (Estimated); Status verified 2013-09

CONDITIONS: HIV Infections
Keywords: HIV-1; Drug Therapy, Combination; Zidovudine; Stavudine; Drug Resistance, Microbial; HIV Protease Inhibitors; CD4 Lymphocyte Count; Ritonavir; Lamivudine; Indinavir; RNA, Viral; Genotype; Reverse Transcriptase Inhibitors; Anti-HIV Agents; Viral Load
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood collection

GROUPS / COHORTS (4):
- 1: Participants who are failing a regimen of ZDV, 3TC, and IDV
- 2: Participants who are failing a regimen of ZDV, 3TC, and SRQ
- 3: Participants who are failing a regimen of ZDV, 3TC, and RTV
- 4: Participants who are failing a regimen of d4T, 3TC, and IDV

SUMMARY:
To determine the short-term virologic and immunologic effects of using plasma genotypic antiretroviral resistance testing (GART) results (interpreted by study virologists AS PER AMENDMENT 9/17/97) in the management of therapy for antiretroviral-experienced patients failing on one of the following regimens:

1. zidovudine (ZDV) + (lamivudine) 3TC + (indinavir) IDV
2. ZDV + 3TC + saquinavir (SQV)
3. ZDV + 3TC + ritonavir (RTV)
4. stavudine (d4T) + 3TC + IDV. [AS PER AMENDMENT 11/26/97: To determine the short-term effects of using plasma GART in the management of antiretroviral-experienced patients failing on a triple drug regimen that includes a single protease inhibitor (indinavir [IDV], saquinavir [SQV], ritonavir [RTV], or nelfinavir [NFV]) and two licensed nucleoside reverse transcriptase inhibitors (NRTIs).] A growing body of evidence suggests that antiretroviral resistance is associated with an increased risk of disease progression and death. All commercially available antiretrovirals and many of those in development have been associated with resistance. Fortunately, techniques are available to define HIV genotypic resistance in "real time" as compared to techniques that measure phenotypic resistance that is not practical in a clinical setting. Using genotypic antiretroviral resistance testing (GART) results, along with other currently available markers, may lead to improved treatment decisions compared with using currently available markers alone.

DETAILED DESCRIPTION:
A growing body of evidence suggests that antiretroviral resistance is associated with an increased risk of disease progression and death. All commercially available antiretrovirals and many of those in development have been associated with resistance. Fortunately, techniques are available to define HIV genotypic resistance in "real time" as compared to techniques that measure phenotypic resistance that is not practical in a clinical setting. Using genotypic antiretroviral resistance testing (GART) results, along with other currently available markers, may lead to improved treatment decisions compared with using currently available markers alone.

128 patients are randomized to GART or no GART within each of four strata defined by current antiretroviral regimen:

1. ZDV plus 3TC plus IDV
2. ZDV plus 3TC plus SQV
3. ZDV plus 3TC plus RTV
4. d4T plus 3TC plus IDV. Each of the four strata contains 22 patients with CD4+ counts of 50 - 199/mm3 and 11 patients with CD4+ counts of 200 - 500/mm3. Upon randomization, clinicians determine a treatment strategy with supplied baseline GART results (GART arm) or without them (no-GART arm). All patients remain on the triple antiretroviral regimen initiated at the randomization visit until at least the 8-week visit. At this time, changes in treatment will be allowed based on an inadequate response to therapy.

[AS PER AMENDMENT 9/17/97: 128 patients are randomized to therapy based on GART results or therapy not based on these results. Patients are stratified into 8 groups defined by current antiretroviral regimen (ZDV/3TC/IDV vs. ZDV/3TC/SQV vs. ZDV/3TC/RTV vs. d4T/3TC/IDV) and screening CD4+ count (50-199 vs. 200-500). Management of patients assigned to the GART group is based on recommendations of study virologists after independent review of patient plasma GART results in addition to current clinical practice. Up to four different treatment regimens using only licensed drugs may be recommended, ranked but considered approximately therapeutically equivalent. The management of patients assigned to the no-GART group is based on current clinical practice and includes only licensed antiretrovirals.] [AS PER AMENDMENT 11/26/97: 160 patients are randomized to GART or no GART within each of 8 strata defined by current antiretroviral regimen (NRTI-1 plus NRTI-2 plus IDV vs. NRTI-1 plus NRTI-2 plus SQV vs. NRTI-1 plus NRTI-2 plus RTV vs. NRTI-1 plus NRTI-2 plus NFV) and screening CD4+ cell count.]

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Documentation of a CD4+ cell count between 50 and 500/mm3 prior to the baseline visit [within 6 weeks prior to baseline visit AS PER AMENDMENT 9/17/97].
* Documentation of either a plasma HIV RNA > 50,000 copies/ml by the Roche Amplicor HIV-1 assay or > 25,000 copies/ml by the Chiron bDNA assay, performed within 30 days prior to the baseline visit. [AS PER AMENDMENT 9/17/97: Documentation of either a plasma HIV RNA level >20,000 copies/ml by the Roche Amplicor HIV-1 assay or >10,000 copies/ml by the Chiron bDNA assay, performed within 6 weeks prior to baseline visit.]
* Documentation of a 3-fold rise in plasma HIV RNA level (using the same assay) or a previously documented plasma HIV RNA at an undetectable level while on the current antiretroviral regimen. [AS PER AMENDMENT 9/17/97: Documentation that the screening plasma HIV RNA level is a 3-fold rise from a previous determination (using the same assay) or documentation of a previous plasma HIV RNA <500 copies/ml while on the current antiretroviral regimen.]
* Signed, informed consent from a parent or legal guardian for patients < 18 years of age.

Prior Medication: Included:

* At least an 18-month cumulative history of antiretroviral therapy [AS PER AMENDMENT 9/17/97: At least a 12-month cumulative history of antiretroviral therapy].

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions are excluded:

* Intercurrent illness (which in the clinician's judgment could influence the HIV RNA level) within 2 weeks prior to, or since, obtaining blood for the screening HIV RNA measurement [within 2 weeks prior to obtaining screening HIV RNA specimen or within 2 weeks prior to baseline visit AS PER AMENDMENT 11/26/97].
* Unwillingness or inability to change antiretroviral therapy.
* Unwillingness to wait up to 30 days after the GART baseline visit to change current triple treatment therapy regimen [AS PER AMENDMENT 9/17/97: Unwillingness to wait until baseline plasma GART results are available to change the current triple therapy regimen].
* Accessibility to previous genotypic or phenotypic resistance testing results.
* Co-enrollment in a clinical trial with anti-HIV drugs.

Concurrent Medication:

Excluded:

* Agents with anti-HIV activity.
* Initiation of treatment with IL-2, interferon, or adefovir dipivoxil.
* Anti-influenza or other vaccines.

Prior Medication:

Excluded:

[AS PER AMENDMENT 11/26/97:

* Use of immunomodulators within 2 weeks prior to obtaining the screening plasma HIV RNA specimen or within 2 weeks prior to the baseline visit.
* Use of any anti-HIV agents, other than drugs in the qualifying triple antiretroviral regimen, within the past 16 weeks.]

Patients must currently be on one of the following triple antiretroviral regimens for at least 16 weeks:

* ZDV + 3TC + IDV
* ZDV + 3TC + SQV
* ZDV + 3TC + RTV
* d4T + 3TC + IDV. [AS PER AMENDMENT 11/26/97: Patients must currently be on a triple antiretroviral regimen that includes a single protease inhibitor (IDV, SQV, RTV, or NFV) and two licensed NRTIs for at least 16 weeks.]

Concurent Treatment: Excluded:

* Vaccination within 2 weeks prior to, or since, obtaining blood for the screening HIV RNA measurement [within 2 weeks prior to obtaining screening plasma HIV RNA specimen or within 2 weeks prior to the baseline visit AS PER AMENDMENT 11/26/97].

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HIV-infected participants currently failing their antiretroviral regimens
Sampling Method: Non-Probability Sample
Enrollment: 148 (Actual)
Dates: Start 1997-08; Primary Completion 1999-01 (Actual); Study Completion 1999-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Baxter J, Study Chair; Mayers D, Study Chair; Merigan T, Study Chair
Locations (24):
- United States (24):
  - Community Consortium / UCSF, San Francisco, California
  - Community Consortium of San Francisco, San Francisco, California
  - Alpine Family Medicine / Janowski, Denver, Colorado
  - Denver CPCRA / Denver Public Hlth, Denver, Colorado
  - S Denver Infectious Diseases Specialists, Denver, Colorado
  - VA Med Ctr, Denver, Colorado
  - Montgomery County Health Dept, Washington D.C., District of Columbia
  - Veterans Administration Med Ctr / Regional AIDS Program, Washington D.C., District of Columbia
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - AIDS Research Alliance - Chicago, Chicago, Illinois
  - Louisiana Comm AIDS Rsch Prog / Tulane Univ Med, New Orleans, Louisiana
  - Wayne State Univ / WSU / DMC HIV / AIDS Program, Detroit, Michigan
  - Henry Ford Hosp, Detroit, Michigan
  - Mercer Area Early Intervention Services, Camden, New Jersey
  - Southern New Jersey AIDS Cln Trials / Dept of Med, Camden, New Jersey
  - North Jersey Community Research Initiative, Newark, New Jersey
  - Partners in Research / New Mexico, Albuquerque, New Mexico
  - Partners Research, Albuquerque, New Mexico
  - T A Ferrill Regional HIV Clinic, Albuquerque, New Mexico
  - Harlem AIDS Treatment Group / Harlem Hosp Ctr, New York, New York
  - The Research and Education Group, Portland, Oregon
  - Philadelphia FIGHT, Philadelphia, Pennsylvania
  - Saint Joseph's Hosp, Philadelphia, Pennsylvania
  - Richmond AIDS Consortium, Richmond, Virginia

REFERENCES:
- [Background] Winters MA, Baxter JD, Mayers DL, Wentworth DN, Hoover ML, Neaton JD, Merigan TC. Frequency of antiretroviral drug resistance mutations in HIV-1 strains from patients failing triple drug regimens. The Terry Beirn Community Programs for Clinical Research on AIDS. Antivir Ther. 2000 Mar;5(1):57-63. PMID 10846594
- [Background] Mayers D. A Pilot Study of the Short-Term Effects of Antiretroviral Management Based on Plasma Genotypic Antiretroviral Resistance Testing (GART) Compared With Antiretroviral Management Without Plasma GART. (abstract no.124)
- [Background] Baxter JD, Mayers DL, Wentworth DN, Neaton JD, Merigan TC. A pilot study of the short-term effects of antiretroviral management based on plasma genotypic antiretroviral resistance testing (GART) in patients failing antiretroviral therapy. Conf Retroviruses Opportunistic Infect. 1999 Jan 31-Feb 4;6th:206 (abstract no LB8)
- [Background] Baxter JD, Mayers DL, Wentworth DN, Neaton JD, Hoover ML, Winters MA, Mannheimer SB, Thompson MA, Abrams DI, Brizz BJ, Ioannidis JP, Merigan TC. A randomized study of antiretroviral management based on plasma genotypic antiretroviral resistance testing in patients failing therapy. CPCRA 046 Study Team for the Terry Beirn Community Programs for Clinical Research on AIDS. AIDS. 2000 Jun 16;14(9):F83-93. doi: 10.1097/00002030-200006160-00001. PMID 10894268
- [Background] Baxter JD, Merigan TC, Wentworth DN, Neaton JD, Hoover ML, Hoetelmans RM, Piscitelli SC, Verbiest WH, Mayers DL; CPCRA 046 Study Team for the Terry Beirn Community Programs for Clinical Research on AIDS. Both baseline HIV-1 drug resistance and antiretroviral drug levels are associated with short-term virologic responses to salvage therapy. AIDS. 2002 May 24;16(8):1131-8. doi: 10.1097/00002030-200205240-00006. PMID 12004271